CLINICAL TRIAL: NCT05737277
Title: Bifidobacterium Adolescentis PRL2019 in Pediatric Irritable Bowel Siyndrome: a Randomized Controlled Trial
Brief Title: Gabapral in Pediatric IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Principal Investigator, Dr. Enrico Felici, Doctor, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAB-IBSPED
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Bifidobacterium Adolescentis PRL2019; IBS; Pediatric

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GABAPRAL (Experimental): Children with irritative bowel sindrome who received 20 Mld UFC of Bifidobacterium adolescentis PRL 2019 once a day for 12 weeks
  Interventions: Drug: Gabapral
- Placebo (Placebo Comparator): Children with irritative bowel sindrome who received placebo once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapral — This will be a randomised, double-blind, placebo-controlled, parallel-arm trial, designed to evaluate the efficacy and safety of Bifidobacterium adolescentis PRL2019 in pediatric patients (> 4 years) with IBS (as assessed according to the Rome IV diagnostic criteria for IBS).
  The study will include a 2-week screening period, and a 12-week placebo-controlled treatment period (Figure 1). After the screening phase, eligible patients will be randomly assigned to either 1 stick containing 20 Mld UFC of Bifidobacterium adolescentis PRL2019 (Gabapral, Pontenure, Italy), or the equivalent placebo once a day, in a 1:1 ratio, for 12 weeks. Study visits will be conducted every 4 weeks during the treatment period.
  Arms: GABAPRAL
Drug: Placebo — This will be a randomised, double-blind, placebo-controlled, parallel-arm trial, designed to evaluate the efficacy and safety of Bifidobacterium adolescentis PRL2019 in pediatric patients (> 4 years) with IBS (as assessed according to the Rome IV diagnostic criteria for IBS).
  The study will include a 2-week screening period, and a 12-week placebo-controlled treatment period (Figure 1). After the screening phase, eligible patients will be randomly assigned to either 1 stick containing 20 Mld UFC of Bifidobacterium adolescentis PRL2019 (Gabapral, Pontenure, Italy), or the equivalent placebo once a day, in a 1:1 ratio, for 12 weeks. Study visits will be conducted every 4 weeks during the treatment period
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a functional gastrointestinal (GI) disorder (FGID) characterized by recurrent episodes of defecation related abdominal pain associated with abnormal bowel habit. Several studies have reported significant alterations in the gut microbiota that may promote the development and persistence of IBS. Some Bifidobacterium species, mainly Bifidobacterium adolescentis, have a documented immunomodulatory effect and can modulate visceral hypersensitivity or improve the integrity of the intestinal epithelium barrier thorough its well-known ability to produce g-aminobutyric acid

Thus, designed a randomised, double-blind, placebo-controlled, parallel-arm study evaluating the efficacy and safety of Bifidobacterium adolescentis PRL2019 on abdominal pain symptoms in pediatric patients with Irritative bowel sindorom

DETAILED DESCRIPTION:
This will be a randomised, double-blind, placebo-controlled, parallel-arm trial, designed to evaluate the efficacy and safety of Bifidobacterium adolescentis PRL2019 in pediatric patients (> 4 years) with Irritative bpwel sindrome (as assessed according to the Rome IV diagnostic criteria for IBS).

The study will include a 2-week screening period, and a 12-week placebo-controlled treatment period. After the screening phase, eligible patients will be randomly assigned to either 1 stick containing 20 Mld UFC of Bifidobacterium adolescentis PRL2019 (Gabapral, Pontenure, Italy), or the equivalent placebo (without the active treatment, once a day, in a 1:1 ratio, for 12 weeks. Study visits will be conducted every 4 weeks during the treatment period. All the subjects will be blindly allocated by means of scratch cards to one of the two treatment groups according to a computer-generated randomisation list provided by our statistician. A validated program will be used by an independent statistician to generate a randomisation list with blocks, block size = 4, pre-allocated to centres. Patients and study investigators will be blinded to the randomisation codes. The codes will be kept confidential until the end of the study when the randomisation code will be broken after the database lock.

All subjects will undergo a formal clinical assessment and will be further phenotyped using validated questionnaires. Number of bowel movements per day and/or week and bowel habit characteristics, will be assessed by the Bristol stool scale.

The protocol will be approved by an independent ethics committee and conducted according to the Declaration of Helsinki and the principles of good clinical practice. The trial will be registered in a public registry.

The primary outcome will be the change in the abdominal pain symptoms (frequency and severity) according to validated score from baseline to the end of the treatment period. Secondary outcomes will be modifications of bowel habits and safety.

Study patients

Eligible patients with symptoms meeting Rome IV criteria for diagnosis of Irritative bowel sindrome will be recruited from Sant'Andrea University Hospital.

Inclusion criteria will comprise a positive diagnosis of all Irritative Bowel Sindrome subtypes, at least 4 and no more of 17 years of age, negative fecal calprotectine and anti-transglutaminasi antibodies.

Exclusion criteria will include the current use of nonsteroidal anti-inflammatory drugs, corticosteroids and mast cell stabilisers, the use of topical or systemic antibiotics in the last month, or the continuous use of stimulant laxatives, major abdominal surgery, inflammatory bowel disease, infectious diarrhoea, allergic diseases and other organic or psychiatric disorders.

Statistical Analysis

The estimated total sample size that was aimed was 96 (48 children per arm) with the power of 80% (alpha of 5%). We estimated a dropout rate of 20% and aimed to recruit 120 participants to provide at least 96 evaluable assessments.

Difference between continuous variables will be assessed either by two-tailed Student t test for values with normal distribution or the MannWhitney test for non-normally distributed variables.

paired samples, based on distribution, Student t test for paired samples or Wilcoxon test will be used. To compare categorical variables chi squared test will be used. The difference between study groups will be considered significant when the P value will be <0.05. Statistical analysis will be performed by using the computer software SPSS 25.0

ELIGIBILITY:
Inclusion Criteria

* IBS subtypes 4 -17 years of age,
* negative fecal calprotectine
* negative anti-transglutaminasi antibodies.

Exclusion Criteria:

* the current use of nonsteroidal anti-inflammatory drugs, corticosteroids and mast cell stabilisers,
* the use of topical or systemic antibiotics in the last month,
* use of stimulant laxatives,
* major abdominal surgery,
* inflammatory bowel disease,
* infectious diarrhoea,
* allergic diseases a
* psychiatric disorders.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Rome IV criteria | 2 months
  The primary outcome will be the improve in the abdominal pain symptoms (frequency and severity) according to validated score from baseline to the end of the treatment period.

SECONDARY OUTCOMES:
bristol stool scale | 6 months
  Secondary outcomes will be modifications of bowel habits and safety.

IPD SHARING:
Plan to Share IPD: Undecided